CLINICAL TRIAL: NCT05395585
Title: The Effect of Placental Spontaneous Delivery Versus Manual Removal on Blood Loss During Cesarean Section. A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MS 290/2022
Record Dates: First submitted 2022-05-25; First posted 2022-05-27 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spontaneous separation (No Intervention)
- Manual separation (Experimental)
  Interventions: Procedure: Manual placental separation

INTERVENTIONS:
Procedure: Manual placental separation — Manual separation of the placenta from uterus
  Arms: Manual separation

SUMMARY:
The mode of placental delivery may contribute to an increase or decrease in the morbidity associated with CS, and many studies have shown it to be a key role in determining the blood loss during CS. Manual removal of the placenta has been implicated in increased blood loss during CS. However, other researchers concluded that it had no detrimental effect on blood loss

ELIGIBILITY:
Inclusion Criteria:

* Age (18 - 35) years.
* Primigravida.
* Unscarred uterus.
* Singleton pregnancy.
* Living baby.
* Body mass index (18 - 30) 37-40 weeks

Exclusion Criteria:

* Emergency cesarean section due to possibility of maternal distress and blood loss.
* Cesarean hysterectomy as the placenta will be removed with the uterus.
* Abnormally adherent placenta: Placenta accrete, percreta or placenta previa due to failure of placental separation.
* Previous cesarean section as the previous scar may affect placental separation.
* Body mass index less than 18 and more than 30 as extremes of body weight may be associated with increased risks of anemia, bleeding and/or infection.
* Suspected chorioamnionitis to decrease the risk of disseminated infection.
* Bleeding disorders to decrease blood loss.
* Multiple pregnancy due to larger placental volume and blood loss compared with singleton.
* Any pelvic surgery (Appendix - Ovarian cyst. - Ectopic Pregnancy - pelvic abscess)
* Women with medical illness e.g. pre-eclampsia, anemia (Hb less than 11 gm/dl), DM, Cardiac, Renal …etc. to decrease the risk of maternal morbidity.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-08 (Actual)

PRIMARY OUTCOMES:
Blood loss | 24 hours
  The blood loss during cesarean section and in the first 24 hours postoperatively will be assessed in a standard manner. Blood will be measured after suction of the mount of amniotic fluid in a separate suction bottle. Amount of blood which collected from towels will be measured according to gravimetric method which reported by Liu et al. (2020).
  - EBV x (Hi-Hf)/Hi: Where the Hi is the preoperative blood hematocrit, Hf is the postoperative one and EBV is the estimated blood volume. The estimated blood volume could be calculated by multiplying weight times average blood volume which is around 65 ml/kg in females (Miller et al., 2000).

CONTACTS AND LOCATIONS:
Overall Officials: Maii Nawara, Study Director — Ain Shams University
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Cairo/القاهرة, Egypt

IPD SHARING:
Plan to Share IPD: Yes